CLINICAL TRIAL: NCT00879177
Title: Contingency Management for Initiating Smoking Abstinence in Patients With Hypertension
Brief Title: Smoking Study With Behavioral Therapy for Hypertensive Patients
Acronym: VANQUISH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, William B. White, Professor of Medicine, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-218; R01DA024667 (NIH)
Record Dates: First submitted 2009-03-24; First posted 2009-04-09 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Cigarette Smoking; Hypertension
Keywords: smoking; varenicline; behavioral therapy; ABPM; hypertension
MeSH Terms: conditions — Cigarette Smoking; Hypertension; Smoking | interventions — Varenicline; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Study drug (varenicline) for 12 weeks, brief smoking cessation counseling for 5 weeks, and ambulatory blood pressure monitoring at Weeks 6 and 24.
  Interventions: Drug: Varenicline
- Group B (Experimental): Study drug (varenicline) for 12 weeks, brief smoking cessation counseling for 5 weeks, ambulatory blood pressure monitoring at Weeks 6 and 24, and behavioral therapy for Weeks 2-5.
  Interventions: Drug: Varenicline; Behavioral: behavioral therapy

INTERVENTIONS:
Drug: Varenicline — Varenicline: 1 tab 0.5mg once a day for 3 days; 1 tab 0.5mg twice a day for 4 days; followed by 1 tab 1mg twice a day for 11 weeks.
  Other Names: CHANTIX
Behavioral: behavioral therapy — confirmed negative smoking status at different time points
  Arms: Group B

SUMMARY:
In total, 260 patients with pre- and stage I hypertension, who are regular smokers, will be randomized to: varenicline alone or varenicline plus behavioral therapy. Patients in both conditions will receive varenicline (titrated to a maximal dose of 1.0 mg twice daily) for 12 weeks along with standard smoking cessation therapy and regular carbon monoxide (CO) and cotinine monitoring. A significantly higher proportion of behavioral therapy patients are expected to achieve and maintain long durations of abstinence than patients receiving varenicline alone. Clinic and 24-hour blood pressure (BP) and heart rate (HR) will be primary clinical outcomes. The investigators expect that BP and HR will decrease more among behavioral therapy than non-behavioral therapy patients and reductions in smoking may mediate decreases in these indices.

ELIGIBILITY:
Inclusion Criteria:

* regular smokers, with no period of abstinence exceeding 3 months in past year
* expired CO of at least 8 ppm
* self-reported desire to stop smoking
* at least 18 years of age
* resting systolic BP of 120-160 mmHg and/or diastolic BP of 80-100 mmHg but otherwise in good health (see exclusion criteria)
* if on antihypertensive medication, have not changed medications during the previous month and do not intend to change in the next 3 months
* English speaking

Exclusion Criteria:

* receipt of smoking cessation treatment (behavioral or pharmacological) in the past month
* serious or unstable medical disease within the past 6 months, including myocardial infarction, cancer, congestive heart failure, kidney failure, stroke, or seizures
* evidence or history of allergic reactions contraindicating varenicline use or clinically significant laboratory or electrocardiographic (ECG) abnormalities
* breastfeeding, pregnant or not using effective contraception if a woman of childbearing potential
* arm circumference of >42 cm, which precludes accurate BP monitoring
* serious psychiatric illness in past 6 months (e.g., schizophrenia, psychosis, suicide risk, drug or alcohol dependence other than nicotine)
* use of tobacco containing products other than cigarettes in past month and do not agree to abstain from use of these products during study participation
* ongoing use of any of the following medications: nicotine replacement therapies, monoamine oxidase inhibitors, antipsychotics, mood stabilizers, or naltrexone
* in recovery for pathological gambling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2009-04; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Short-term and long-term smoking abstinence and improved health benefits | Weeks 5,6,8,12,24,36,52

SECONDARY OUTCOMES:
Decrease in blood pressure and heart rate in hypertensive subjects | Week 6 and Week 24

CONTACTS AND LOCATIONS:
Overall Officials: William B White, M.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No